CLINICAL TRIAL: NCT04684316
Title: Economic Evaluation of an Online Screening Tool With Selective Follow-up Versus Periodic Health Screening by the Occupational Physician
Brief Title: Economic Evaluation of Periodic Occupational Health Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Belgian Association for Occupational Physicians (Unknown); IDEWE Occupational Health Services (Other); Liantis (Unknown); Mensura (Unknown)
Responsible Party: Principal Investigator, Jeroen Luyten, Associate professor of health economics, KU Leuven
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: EZG-D7685
Record Dates: First submitted 2020-12-10; First posted 2020-12-24 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Occupational Health; Screening; Surveys and Questionnaires
Keywords: occupational medicine; survey; periodic health surveillance

STUDY DESIGN:
Intervention Model Description: Employees within the same hospital are prospectively and randomly allocated to one of two groups: an intervention group receives an electronic survey with selective follow-up by the occupational physician, and a control group where all employees undergo a periodic health screening by the occupational physician. The survey is thus used as part of the intervention, as an algorithm (based on a scoring system of the survey) which determines who should be seen by the occupational physician is evaluated. However, the survey is also used to gather data on how the selective referral affects outcomes. There are three measurement moments (each time with the same survey, and in both groups). First, baseline outcomes are measured in June 2019, after which selective follow-up in the intervention group and contact with the OP in the control group is organised in June-December 2019. Differences in outcomes between groups are then measured in February 2020, and in September 2020.
Who Masked: Participant
Masking Description: Participants are partially masked: if a participant is invited for a consultation with the occupational physician, they do not know whether this is because they are in the control group, or because they were in the intervention group and selected on the basis of their scores. Participants that do not see the occupational physician can deduce that they are part of the intervention group. Care providers, investigators, and outcomes assessors know to which group an individual pertains as this is required for the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care-as-usual: all consult physician (No Intervention): All employees at risk are invited to attend screening. Upon arrival, several biometrics are measured (weight, length, Body Mass Index, blood pressure), along with spirometries, a vision test, and a blood and urine test. The OP then investigates the general health status and systems of the employee, which includes an anamnesis with questions about new health burdens or changes in occupational risks, follow-up questions on previous complaints, medical advice, referral to a healthcare provider, or booking another appointment with an occupational health specialist. After the PHS, a (employee-unique) link to an online questionnaire is sent by email to gather information on final (health, health care use, absenteeism and presenteeism) and intermediary (health literacy, help-seeking behaviour) outcomes.
- Intervention: Electronic survey with selective consultations (Experimental): In the intervention group, all employees at risk receive a (employee-unique) link to an online health screening questionnaire by email. Dependent upon their answers, 20% of the employees (i.e. the 20% of the employees that mostly need contact with the OP) are referred to the occupational physician for a discussion of the results. The OP then gives medical advice, refers to a healthcare provider (e.g. general practitioner or specialist), or books a (follow-up) appointment with an occupational health specialist (OP, occupational nurse, etc.).
  Interventions: Other: Electronic survey with selective consultations

INTERVENTIONS:
Other: Electronic survey with selective consultations — Participants complete an online questionnaire, after which the 20% employees that mostly need contact with the occupational physician (based on their survey score) are invited to a consultation with the occupational physician.
  Arms: Intervention: Electronic survey with selective consultations

SUMMARY:
In Belgium, Periodic Health Screenings (PHS) are obliged by law for several occupations, including safety functions, jobs with heightened vigilance, work that involves physical, biological or chemical agents or tasks that are an ergonomic or mental burden. Scientifically it remains an open question whether these screenings guarantee the prevention of later health problems or problems with functioning at work.

The objective of this study is to compare the cost-effectiveness of PHS with an online health screening tool with selective follow-up. In five Flemish hospitals, the employees eligible for PHS (exempting frequent exposure to ionizing radiation, preparation of cytostatics, or exposure to carcinogens, mutagens, or reprotoxic substances) are randomly assigned to a control group (receiving classical PHS at the occupational physician), or an intervention group (e-tool with selective follow-up by the physician). In the intervention group, 20% of the employees is seen by the occupational physician, based on their responses to the questionnaire. The intervention- and control group complete the questionnaire three times: before the study start (June 2019), in February 2020, and in September 2020. The study ends in March 2021.

The survey is developed as part of the study. On the one hand it contains questions for the cost-effectiveness analysis: health care use, absenteeism and presenteeism, and health literacy. On the other hand, a validated questionnaire is developed based on a systematic review of existing validated and reliable instruments, a Delphi panel of occupational physicians, and a pilot- and field study that test the reliability and validity of the survey (and its referral to the occupational physician). For the latter, the employees' health, occupational risks, work ability, and lifestyle (alcohol abuse, drug abuse, physical activity, and nutrition) are surveyed. Access to the occupational physician remains guaranteed by means of an additional question ("Do you wish to discuss the results of your survey with the occupational physician?") and as spontaneous consultations with the occupational physicians remain possible before, during, and after the trial.

The survey platform Qualtrics is used for data collection. Researchers have no insight in personal data, nor the medical files of employees, and only analyse the coded data from the surveys. Invitations for the survey are sent by the occupational physician. The coded questionnaires are saved on a KU Leuven survey, following the ISO-9001-procedure and the legal data storage period. The employer has no insight in the data. The study is performed by Jonas Steel, supervised by prof. dr. Jeroen Luyten and prof. dr. Lode Godderis, and financed by the Belgian Association for Occupational Physicians, and three external services for prevention and protection at work: IDEWE, Liantis, and Mensura.

DETAILED DESCRIPTION:
In Belgium, Periodic Health Screenings (PHS) are obliged by law for several occupations and allow for early detection of health problems, advice towards risk-free behaviour, timely risk reductions or referrals to other care personnel. This makes them one of the key preventive activities of the occupational physician (OP). However, there are as of yet no strong research indications for the optimal organisation of these occupational health screenings. A recent systematic review of general health screening (not only at the workplace) did not find studies that indicated an effect (e.g. on general mortality, cardiovascular mortality, or cancer mortality), but indicated they could lead to adverse effects such as overtreatment or misplaced reassurance. Reviews in other domains such as vision screening of older drivers, tuberculosis screening of healthcare workers, tomography for lung cancer, of pre-employment investigations frequently found too few high quality studies to draw strong conclusions. There is some evidence for the effectiveness of biometric screening in reducing the number of non-communicable diseases, especially when aimed at higher risk employees or if they are combined with well-designed health programmes. However, it remains an open question whether more focused occupational screenings with risk-selection, as is the case in Belgium and the Netherlands, are beneficial.

This protocol will therefore present a study on annual periodic health screenings (PHS). In this sense, it will contribute to evidence-based decision-making for policy makers, who are currently planning to change the legislation.

A theoretically ideal experiment would compare a group of employees undergoing periodic health screening with a group without an intervention. However, three factors make the formulation of an alternative intervention necessary. Firstly, from an ethical point of view, adequate medical follow-up should be provided for all participants in the study. Secondly, current legislation requires employees to undergo screening for "risky" occupational activities to assess their aptitude for those activities. Thirdly, it is important to provide employers with an alternative form of care or follow-up, since it would not be beneficial (for any party) if employers paid the same fees to the Services for Prevention and Protection at Work (SPPW), but got less care in return. The experiment will therefore compare care-as-usual (periodic health screenings by the OP - the control group) with employees that complete an electronic health survey with selective follow-up (the intervention group). The latter encompasses that the employees' answers on the health screening tool determine whether he/she will be seen by the OP. This allows immediate data collection for the experiment, and at the same time guarantees follow-up of employees with health problems by SPPW.

The survey wants to answer to the demands (of a good PHS) of the International Labour Office by focusing on primary (sometimes secondary) prevention, by taking a risk analysis as a starting point, by allowing for both individual and collective measures, by formulating goals in advance, and because finding problems leads to adequate action. To fulfil these goals, the questionnaire will not only make use of health information (health status, early detection of occupational disease, accidents), but also of other signals that could point towards a higher risk of absence or reduced functioning: absenteeism, presenteeism, health care use, working conditions, job-specific factors, and lifestyle. In addition, the health literacy of personnel is taken into account to assess how well information about health at work (eg coming from the OP) is understood. Briefly summarized, health literacy contains three dimensions: access - how employees are able to seek and obtain health information - "understanding" - the expectations, perceived utility and interpretation of health information - and "behaviour" - the employee's intention to change behaviour as well as his behaviour itself. Finally, it is possible to measure the help-seeking behaviour of employees, to assess their tendency to seek medical care when needed. By incorporating these aspects into the survey and study, we will circumvent the complication that many preventive interventions have to face: health ameliorations and decreases in health care use, absenteeism and presenteeism only occur after several years.

ELIGIBILITY:
Inclusion Criteria:

* all personnel types that are eligible for periodic health screenings: personnel with safety functions, jobs with heightened vigilance, work that involves physical, biological or chemical agents or tasks that are an ergonomic or mental burden
* working age (18-70 years old)
* able to understand and answer the questionnaire in Dutch

Exclusion Criteria:

* occupational groups that perform especially risky activities (frequent exposure to ionizing radiation, preparation of cytostatics, or exposure to carcinogens, mutagens, or reprotoxic substances)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 889 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Self-perceived health | change after 15 months
  Self-perceived health using a visual analog score: 0-100 (from worst health the employee can imagine to the best health the employee can imagine)
Incidence of musculoskeletal health functioning problems | change after 15 months
  Count of how many respondents indicated to have musculoskeletal health functioning problems
Stress | change after 15 months
  Score that represents the risk of stress based on the Copenhagen Psychosocial Questionnaire: 0-12 (from low to high risk of stress)
Burnout | change after 15 months
  Score that represents the risk of burnout based on the Copenhagen Psychosocial Questionnaire: 0-16 (from low to high risk of burnout)
Sleep problems | change after 15 months
  Score that represents the risk of sleep problems based on the Copenhagen Psychosocial Questionnaire: 0-16 (from low to high risk of burnout)
General mental health | change after 15 months
  Score that represents the general mental health based on the General Health Questionnaire: 0-12 (from worst to best mental health)
Need for recovery after work | change after 15 months
  Score that represents the need for recovery after work, based on the Need for Recovery scale: 0-11 (from lowest to highest need for recovery after work)
Absenteeism | change after 15 months
  Absenteeism in days absent using the IMTA Productivity Cost Questionnaire (iPCQ)
Presenteeism | change after 15 months
  Presenteeism using the IMTA Productivity Cost Questionnaire (iPCQ), which uses a visual analog score to indicate how much work the employee could perform compared to a normal working day
Spontaneous consultations with the occupational physician | change after 15 months
  Self-reported number of spontaneous consultations the employee had with the occupational physician
Referrals to other health providers | change after 15 months
  Number of contact moments with other healthcare providers based on a referral by the occupational physician

SECONDARY OUTCOMES:
Health literacy | change after 15 months
  Score representing the health literacy of the employee, based on an adapted version of the European Health Literacy Survey (EU-HLS): 0-64 (low to high health literacy)
Help-seeking behaviour | change after 15 months
  Score representing the help-seeking behaviour of the employee, based on the General Help-Seeking Questionnaire: 0-128 (high self-assessed probability of seeking help to low self-assessed probability of seeking help)

CONTACTS AND LOCATIONS:
Overall Officials: Jonas S Steel, Msc, Principal Investigator — KU Leuven
Locations (4):
- Belgium (4):
  - Heilig Hart Leuven, Leuven, Flanders
  - AZ Nikolaas, Sint-Niklaas, Flanders
  - Heilig Hart Tienen, Tienen, Flanders
  - AZ Vesalius, Tongeren, Flanders

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive medical nature of the data, no data will be shared with other researchers.

REFERENCES:
- [Background] Krogsboll LT, Jorgensen KJ, Gotzsche PC. General health checks in adults for reducing morbidity and mortality from disease. Cochrane Database Syst Rev. 2019 Jan 31;1(1):CD009009. doi: 10.1002/14651858.CD009009.pub3. PMID 30699470
- [Background] Larsen AK, Holtermann A, Mortensen OS, Punnett L, Rod MH, Jorgensen MB. Organizing workplace health literacy to reduce musculoskeletal pain and consequences. BMC Nurs. 2015 Sep 17;14:46. doi: 10.1186/s12912-015-0096-4. eCollection 2015. PMID 26388697
- [Background] Sorensen K, Van den Broucke S, Fullam J, Doyle G, Pelikan J, Slonska Z, Brand H; (HLS-EU) Consortium Health Literacy Project European. Health literacy and public health: a systematic review and integration of definitions and models. BMC Public Health. 2012 Jan 25;12:80. doi: 10.1186/1471-2458-12-80. PMID 22276600